CLINICAL TRIAL: NCT07396805
Title: A Randomized Controlled Trial of Food Is Medicine Approaches for Obesity Treatment in Adults With Food Insecurity
Brief Title: Trial of Food Is Medicine Approaches for Obesity Treatment in Adults With Food Insecurity
Acronym: EatWell Rx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00528955; R01NR021699 (NIH)
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
Keywords: obesity; weight loss; food insecurity; nutrition
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BWL-Alone (Active Comparator): Participants receive BWL-Alone
  Interventions: Behavioral: BWL
- BWL+Voucher (Experimental): Participants receive BWL+Voucher
  Interventions: Behavioral: BWL; Other: VOUCHER
- BWL+Home (Experimental): Participants receive BWL+Home
  Interventions: Behavioral: BWL; Other: HOME

INTERVENTIONS:
Behavioral: BWL — Participants will receive a lifestyle modification program consisting of behavioral, physical activity, and dietary counseling delivered over 21, approximately 15 minute sessions delivered by trained interventionists. Sessions will be weekly during weeks 0-4, every other week during weeks 6-24, monthly during weeks 25-52. Treatment will be delivered remotely.
Other: VOUCHER — During the initial 24 weeks, participants randomized to this group will receive the BWL program along with food vouchers distributed in the form of grocery store gift cards. Gift cards worth $60 will be emailed to participants every 2 weeks after their BWL session. From weeks 24-52, participants will continue to have monthly counseling sessions.
  Arms: BWL+Voucher
Other: HOME — During the initial 24 weeks, participants assigned to this group will receive home-delivered, medically tailored groceries alongside BWL. The contents of each box will be approximately $60 ($30/week) and sent using Instacart. From weeks 24-52, participants will continue to have monthly counseling sessions.
  Arms: BWL+Home

SUMMARY:
The goal of this clinical trial is to learn if increased access to healthy foods, combined with behavioral weight loss (BWL) interventions, results in greater weight loss for adults with obesity and food insecurity. It will also learn about changes in health-quality of life and dietary quality. The main questions it aims to answer are:

* Does BWL, combined with either home-delivered, medically-tailored (HOME) groceries or grocery vouchers (VOUCHER), result in greater weight loss than BWL alone?
* Is the addition of HOME to BWL more effective at supporting adults with food insecurity and obesity to lose weight when compared to BWL and VOUCHER?

DETAILED DESCRIPTION:
Participants will:

* Receive 21 sessions of BWL over 52 weeks delivered 1-on-1 with a counselor
* Visit the research team for 4 in-person assessments to assess measures like height, weight, blood pressure, pulse, complete dietary assessments, questionnaires and interviews, and evaluate skin carotenoid levels (a non-invasive measure)
* Be randomized (like picking numbers from a hat) to BWL-Alone; BWL+VOUCHER; or BWL+HOME. Participants in BWL+VOUCHER will receive grocery store gift cards every 2 weeks for the first 24 weeks of the study. Participants in BWL+HOME will receive groceries delivered to the home every 2 weeks for the first 24 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30 kg/m2
* Screening positive for food insecurity using the well-validated, 10-item US Adult Food Security Survey Module.
* Age 18 years and older
* Completion of baseline assessments
* Ability to engage in physical activity (i.e., can walk at least 2 blocks without stopping for rest)
* Willing and able to provide pictures of food receipts to study team (or mail receipts to study team)
* Willing and able to provide written informed consent and participate in all study activities
* Female participants of child-bearing potential must agree in writing to use an approved method of contraception during the study

Exclusion Criteria:

* Significant psychiatric conditions (e.g., active substance abuse, schizophrenia) that may pose a risk to the participant during intervention, cause a change in weight, or limit ability to adhere to the program's behavioral recommendations
* Pregnant or planning pregnancy in the next year
* Planned move from the Baltimore area in the next year
* Recently began a course of or changed the dosage of medication that can cause significant weight change (±5 kg)
* Previous or planned obesity treatment with surgery or a weight-loss device
* Weight loss of >5 kg in the previous 90 days
* Household member already participating in study due to potential contamination effects
* Lack of stable residence and ability to store and prepare food
* Lack of telephone
* Severe food allergies
* Following a specialized dietary regimen (e.g., gluten-free)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Percent initial weight loss at week 24 (BWL+VOUCHER and BWL+HOME to BWL-Alone) | Baseline to 24 weeks
  Comparison of BWL+VOUCHER and BWL+HOME to BWL-Alone for weight loss (percent of baseline weight) at 24 weeks

SECONDARY OUTCOMES:
Percent initial weight loss at week 24 (BWL+VOUCHER versus BWL+HOME) | Baseline to 24 weeks
  Comparison of BWL+VOUCHER versus BWL+HOME for weight loss (percent of baseline weight) at 24 weeks
Percent initial weight loss at week 52 (BWL+VOUCHER and BWL+HOME to BWL-Alone) | Baseline to 52 weeks
  Comparison of BWL+VOUCHER and BWL+HOME to BWL-Alone for weight loss (percent of baseline weight) at 52 weeks
Percent initial weight loss at week 52 (BWL+VOUCHER versus BWL+HOME) | Baseline to 52 weeks
  Comparison of BWL+VOUCHER versus BWL+HOME for weight loss (percent of baseline weight) at 52 weeks
Change from baseline to weeks 24 and 52 in SF-36 Physical Component Score | Baseline to week 24 and week 52
  BWL-Alone, BWL+VOUCHER, and BWL+HOME in changes from baseline to weeks 24 and 52 in SF-36 Physical Component Score. Scores range from 0 (lowest) to 100 (highest/best).
Change from baseline to weeks 24 and 52 in SF-36 Mental Component Score | Baseline to week 24 and week 52
  BWL-Alone, BWL+VOUCHER, and BWL+HOME in changes from baseline to weeks 24 and 52 in SF-36 Mental Component Score. Scores range from 0 (lowest) to 100 (highest/best).
Change from baseline to weeks 24 and 52 in total Impact of Weight on Quality of Life scale | Baseline to week 24 and week 52
  BWL-Alone, BWL+VOUCHER, and BWL+HOME in changes from baseline to weeks 24 and 52 in total Impact of Weight on Quality of Life scale. Scores range from 0 (lowest) to 100 (highest/best).
Change from baseline to weeks 24 and 52 in total Healthy Eating Index score as measured using the Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool | Baseline to week 24 and week 52
  BWL-Alone, BWL+VOUCHER, and BWL+HOME in changes from baseline to weeks 24 and 52 in total Health Eating Index score. Scores range from 0 (lowest) to 100 (highest/best which reflect the set of foods aligns with key dietary recommendations and dietary patterns published in the Dietary Guidelines).
Change from baseline to weeks 24 and 52 in skin carotenoid levels as measured by the Veggie Meter | Baseline to week 24 and week 52
  BWL-Alone, BWL+VOUCHER, and BWL+HOME in changes from baseline to weeks 24 and 52 in skin carotenoid levels with scores ranging from 0 (lowest) to 800 (highest)
Incremental cost-effectiveness per unit decrease in weight (kg) | Baseline to week 24 and week 52
  This measure describes the additional cost required to achieve one kilogram of weight loss with BWL+VOUCHER or BWL+HOME compared with BWL-Alone. It is calculated by dividing the difference in total costs between the two groups by the difference in average weight loss. Lower values indicate that the intervention achieves weight loss at a lower cost.

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Chao, PhD, CRNP, FNP-BC, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States